CLINICAL TRIAL: NCT04135157
Title: Research of the Effects of Pectoralis Nerve Block II and Erector Spina Plan Block in Breast Cancer Surgery
Brief Title: Pectoral Nerve Block II and Erector Spine Plane Block in Breast Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Collaborators: CENGİZ KAYA (ckaya) (Unknown)
Responsible Party: Principal Investigator, Caner Genç, Medical Doctor, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: PA191001001
Record Dates: First submitted 2019-10-19; First posted 2019-10-22 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Anesthesia; Analgesia; Acute Pain; Chronic Pain; Pectoralis Nerve Block; Erector Spine Plane Block; Patient Controlled Analgesia
Keywords: Regional Anesthesia; Acute and chronical pain; Pectoralis nerve block; Erector spine plane block
MeSH Terms: conditions — Agnosia; Acute Pain; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Randomization of the study will be done by a doctor who will not participate in patient follow-up with closed envelopes using computer generated generated random numbers.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The anesthesia doctor who will perform the peripheral nerve block will be informed with a sealed envelope by an independent assistant outside the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PECS II or ESP (Experimental): PECS II or ESP block are performed 30 minutes before general anesthesia. PCA is used for all the patients in the first 24 hours postoperatively.
  Interventions: Procedure: Pectoralis nerve block II; Procedure: Erector spine plane block
- Control (Active Comparator): In the control group, patients will have only general anesthesia. PCA is used for all the patients in the first 24 hours postoperatively.
  Interventions: Other: Control

INTERVENTIONS:
Procedure: Pectoralis nerve block II — PECS II block will be performed 30 min. before general anesthesia.
  Other Names: PECS II
  Arms: PECS II or ESP
Procedure: Erector spine plane block — ESP block will be performed 30 minutes before general anesthesia.
  Other Names: ESP
  Arms: PECS II or ESP
Other: Control — Only general anesthesia will be performed.
  Arms: Control

SUMMARY:
This study evaluates the analgesic effects of pectoralis nerve block (PECS II) and erector spinae plane block (ESP) in patients having segmental mastectomy and sentinel lymph node biopsy (SLNB). Each one-third of patients will have ESP block and pectoralis nerve block (PECS II) 30 min before general anesthesia , while other one-third of patients will have only general anesthesia.

DETAILED DESCRIPTION:
It has been proven that PECS II and ESP both supply effective analgesia in the first 24 hours after mastectomy. But they do so by different mechanishms.

This study is to survey that ESP and PECS II may supply acute and chronic analgesia by reducing pain scores in the first 24 hours and 3 months after the surgery, also the comparison of the analgesic activity among themselves for acute / chronic pain and opioid consumption will be searched.

In this study patients are divided into three groups. Patients in PECS group will have PECS II block in a separate section from the operating rooms (PNB practice room). In addition, patient controlled analgesia (PCA) will be used in the first 24 hours postoperatively.

Patients in ESP group will have ESP block in a separate section from the operating rooms (PNB practice room). In addition, PCA will be used in the first 24 hours postoperatively.

Patients in control group will not be performed nerve block. Only general anesthesia (GA) will be performed in the operation room. In addition, PCA will be used in the first 24 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2 patients between the age of 18-65, scheduled for elective unilateral segmental mastectomy + sentinel lymph node biopsy

Exclusion Criteria:

* Age <18 or> 65, ASA 3-4 patients
* Obesity (> 100 kg, BMI> 35 kg / m2)
* Patients undergoing bilateral mastectomy
* Pregnancy
* Contraindication of regional anesthesia (coagulopathy, abnormal INR, thrombocytopenia, infection at the injection site)
* Serious renal, cardiac, hepatic disease
* Hypersensitivity to local anesthetics or a history of allergy
* Patients with a history of opioid use longer than four weeks
* Patients with psychiatric disorders or communication difficulties
* Patients with chest deformity
* Patients with previous breast surgery except diagnostic biopsies
* Patients who do not want to participate

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with breast cancer having segmental mastectomy and sentinel lymph node biopsy (SLNB)
Enrollment: 90 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Opioid consumption in the first 24 hours after surgery | 1 day
  Morphine consumption in the first 24 hours will be counted by IV PCA. Patients will be able to request opioids via PCA device when the vas score is 4 points or more when the arm is in the resting position.

SECONDARY OUTCOMES:
Post-operative acute pain | 1 day
  Pain status will be evaluated based on VAS scores in two different positions: arm at rest and arm in abduction. Pain status will be evaluated at 1-3-6-12-24. hours after surgery. Each VAS is scores 0-10. (0=no pain ; 10=pain as bad as can be)
Remifentanil consumption during the surgery | During the surgery
  Following induction of general anesthesia, anesthesia maintenance will be continued with sevoflurane to BIS 40-60 (bispectral index). When the BIS is between 40-60, remifentanil infusion rate will be changed considering ± 20% changes in blood pressure compared to baseline values.The total amount of remifentanil consumed will be recorded.
The incidences of post-operative nausea and vomiting (PONV) | 1 day
  The patients will be evaluated according to the five-stage verbal descriptive PONV scale. If it is 3 points or more, ondansetron 4 mg IV will be administered. Wait for 8 hours for the next dose of ondansetron. (0 = None, 1 = Slight nausea, 2 = Moderate nausea, 3 = Once vomiting, 4 = vomiting more than one)
The number of patient required rescue analgesia | 1 day
  The number of patient requires rescue analgesic will be recorded at 1-3-6-12-24. hours after surgery
Post-operative chronic pain | 3. month after surgery
  Pain status will be evaluated in the third month after surgery based on VAS scores in two different positions: arm at rest and arm in abduction. Each VAS is scores 0-10. (0=no pain ; 10=pain as bad as can be)

OTHER OUTCOMES:
The time of first analgesic demand from the PCA device. | 1 day
  The time of first analgesic demand was defined as the time to first PCA bolus after patient PACU arrival.

CONTACTS AND LOCATIONS:
Overall Officials: CENGİZ KAYA, MD, Study Director — Ondokuz Mayıs University Faculty of Medicine
Locations (1):
- Ondokuz Mayıs University Faculty of Medicine, Samsun, Turkey (Türkiye)